CLINICAL TRIAL: NCT05522192
Title: Clinical Study of Venetoclax Combined With Mitoxantrone Liposome in the Treatment of Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Clinical Study of Mitoxantrone Hydrochloride Liposome Injection in Subjects With Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hui Zeng (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Hui Zeng, chief physician, First Affiliated Hospital of Jinan University
Organization: First Affiliated Hospital of Jinan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-AML-K04
Record Dates: First submitted 2022-08-12; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia
Keywords: venetoclax; Mitoxantrone liposomes; Acute myeloid leukemia
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax-Mitoxantrone liposome (Experimental): Phase I
  Mitoxantrone liposome
  * Level 1: 24mg/m^2, ivgtt, d1;
  * Level 2: 30mg/m^2, ivgtt, d1;
  * Level 3: 36mg/m^2, ivgtt, d1;
  Venetoclax: 100mg po d1, 200mg po d2, 400mg po d3-28.
  Every 4 weeks is a cycle, a total of 2 cycles, the first cycle to observe DLT.
  Phase II
  Mitoxantrone liposome: RP2D
  Venetoclax: 100mg po d1, 200mg po d2, 400mg po d3-28.
  28 days is a cycle, and a maximum of 6 cycles can be carried out. If the patient achieves CR, CRi or PR, if the patient can tolerate it, it will be used for 6 cycles; if the patient is suitable for transplantation, it can also enter the transplantation path; If the patient was evaluated as NR (no response) after 2 cycles, he could withdraw from the study.
  Interventions: Drug: Mitoxantrone liposome; Drug: Venetoclax

INTERVENTIONS:
Drug: Mitoxantrone liposome — Phase I: 24mg/m2, 30 mg/m2, 36mg/m2, IV, d1; Phase II: RP2D.
  Other Names: Mitoxantrone Hydrochloride Liposome Injection
Drug: Venetoclax — Phase I/II: 100mg po d1，200mg po d2，400mg po d3-28.
  Other Names: Venclexta

SUMMARY:
This study is an open-label, single-arm, phase I/II clinical study. Phase I is a multi-center, dose-escalation study, aiming to explore the maximum tolerated dose (MTD) of venetoclax combined with mitoxantrone liposome in the treatment of relapsed or refractory acute myeloid leukemia (AML), and determine the recommended dose for phase II (RP2D); Phase II is a multi-center, exploratory study, aiming to explore efficacy of venetoclax combined with mitoxantrone liposome in the treatment of relapsed and refractory AML patients, and to explore the differences in the efficacy of this combination therapy with different gene mutations.

DETAILED DESCRIPTION:
This study is an open-label, single-arm, phase I/II clinical study. Phase I is a multi-center, dose-escalation study. Following the "3+3" principle, it plans to recruit 9-18 patients with clinically diagnosed relapsed or refractory AML who will be treated with venetoclax and mitoxantrone liposome, in order to explore the MTD of mitoxantrone liposome, and determine the RP2D. Mitoxantrone liposome began to explore the dose from 24 mg/m^2, and every 4 weeks (28 days) was a cycle. Three dose groups of 24, 30 and 36 mg/m^2 were preseted; The trial phase includes screening period (within 28 days), treatment period (planned 2 cycles), follow-up period (RFS and OS follow-up, planned 1 year).

Phase II is a multi-center, exploratory study, aiming to explore efficacy of venetoclax combined with mitoxantrone liposome in the treatment of relapsed or refractory AML patients, and to explore the differences in the efficacy of this combination therapy with different gene mutations. After Phase I reaches MTD and the dose of Phase II is determined, Phase II clinical trials will be carried out. The phase II trial phase includes screening period (within 28 days) , treatment period (planned 6 cycles ) and a follow-up period (RFS and OS follow-up, planned for 1 year).

ELIGIBILITY:
Inclusion Criteria:

1. AML confirmed by bone marrow cytology and pathology;
2. Meet the diagnostic criteria for relapsed and refractory AML. Diagnostic criteria for relapsed AML: leukemia cells reappeared in peripheral blood after complete remission or blast cells in bone marrow >0.05 (except for other reasons such as bone marrow regeneration after consolidation chemotherapy) or extramedullary leukemia cell infiltration. Diagnostic criteria for refractory AML: naive patients who were ineffective after 2 courses of standard regimens; patients who relapsed within 12 months after consolidation and intensive therapy after CR; patients who relapsed after 12 months but were ineffective after conventional chemotherapy; 2 or more Secondary relapse; persistent extramedullary leukemia;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2;
4. Liver and kidney function: Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN) (≤5 x ULN for patients with liver infiltrates); Total bilirubin ≤1.5 x ULN (≤3 x ULN for patients with liver infiltration); Serum creatinine ≤1.5 x ULN;
5. Normal cardiac function: left ventricular ejection fraction (LVEF) ≥ 45% assessed by echocardiography or radionuclide active angiography (MUGA);
6. Pulmonary function: dyspnea ≤ CTC AE grade 1 and SaO2 ≥ 92% in indoor air environment;
7. The expected survival time is greater than 3 months;
8. Patients voluntarily participated in this study and signed the informed consent.

Exclusion Criteria:

1. The subject had previously received any of the following anti-tumor treatments: a)Those who have previously received mitoxantrone or mitoxantrone liposome; b)Previously received doxorubicin or other anthracycline treatment, and the total cumulative dose of doxorubicin is more than 360 mg/m^2 (1 mg doxorubicin converted from other anthracycline drugs is equivalent to 2 mg daunorubicin or 0.5 mg idarubicin); c)Have received anti-tumor treatment (including chemotherapy, targeted therapy, hormone therapy, taking traditional Chinese medicine with anti-tumor activity, etc.) or participated in other clinical trials and received clinical trial drugs within 4 weeks before the first use of the study drugs;
2. Heart function and disease meet one of the following conditions: a)Long QTc syndrome or QTc interval > 480 ms; b)Complete left bundle branch block, grade II or III atrioventricular block; c)Serious and uncontrolled arrhythmias requiring drug treatment; d)New York Heart Association grade ≥ II; e)A history of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically serious pericardial disease, or ECG evidence of acute ischemia or active conduction system abnormalities within 6 months before recruitment.
3. Identify patients with central nervous system invasion;
4. Other malignancies, except for effectively controlled non melanoma skin basal cell carcinoma, breast / cervical carcinoma in situ, and other malignancies that have been effectively controlled without treatment in the past five years;
5. Non controlled systemic diseases (such as active infection, non controlled hypertension, diabetes, etc.);
6. Human immunodeficiency virus (HIV) infection (HIV antibody positive);
7. Active hepatitis B and C infection (hepatitis B test: if there is a positive hepatitis B surface antigen or core antibody, add HBV DNA, and the hepatitis B virus DNA exceeds 1x10^3 copies/mL to exclude; hepatitis C: if the hepatitis C antibody is positive, further test HCV RNA, hepatitis C Viral RNA exceeding 1x10^3 copies/mL was excluded);
8. Hypersensitivity to any study drug or its components;
9. Pregnant women, lactating women, patients who refused to take effective contraceptive measures during the study;
10. Serious neurological or psychiatric history;
11. Unsuitable subjects for this study determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Phase I: MTD of mitoxantrone liposomes | At the end of Cycle 1 (each cycle is 28 days)
  To evaluate the tolerability of mitoxantrone liposomes combination regime
Phase II: Composite complete remission rate (CRc) | At the end of Cycle 2 (each cycle is 28 days)
  To evaluate the efficacy of anti-leukemia

SECONDARY OUTCOMES:
Phase I: Composite complete remission rate (CRc) | At the end of Cycle 2 (each cycle is 28 days)
  To evaluate the efficacy of anti-leukemia
Phase I: Objective response rate (ORR) | At the end of Cycle 2 (each cycle is 28 days)
  To evaluate the efficacy of anti-leukemia
Phase I: Relapse free survival (RFS) | Up to 2 years
  To evaluate the efficacy of anti-leukemia
Phase I: Overall survival (OS) | Up to 2 years
  To evaluate the efficacy of anti-leukemia
Phase I: Safety: Hematologic and non-hematologic toxicities (NCI CTCAE v5.0) | From the initiation of the first dose to 28 days after the last dose
  To identify the incidence of AE and SAE in clinical trial
Phase II: Objective response rate (ORR) | At the end of Cycle 2 (each cycle is 28 days)
  To evaluate the efficacy of anti-leukemia
Phase II: Relapse free survival (RFS) | Up to 4 years
  To evaluate the efficacy of anti-leukemia
Phase II: Overall survival (OS) | Up to 4 years
  To evaluate the efficacy of anti-leukemia
Phase II: Safety: Hematologic and non-hematologic toxicities (NCI CTCAE v5.0) | From the initiation of the first dose to 28 days after the last dose
  To identify the incidence of AE and SAE in clinical trial

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zeng, M.D, Principal Investigator — First Affiliated Hospital of Jinan University
Locations (1):
- First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China